CLINICAL TRIAL: NCT04319198
Title: Open-label Rollover Study to Evaluate Long-Term Safety in Subjects With Metastatic Solid Tumors That Are Benefiting From Continuation of Therapy With Sacituzumab Govitecan
Brief Title: Rollover Study in Participants With Metastatic Solid Tumors Benefiting From Therapy With Sacituzumab Govitecan-hziy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-14; 2023-505336-34 (Other: European Medicines Agency)
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Solid Tumors
Keywords: ADC; Antibody-Drug Conjugate; Trop-2; SN-38
MeSH Terms: interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) (Experimental): All participants who previously received SG in the parent study (IMMU-132-01) will continue to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until progressive disease (PD), toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
  Interventions: Drug: Sacituzumab Govitecan-hiy
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) (Experimental): All participants who previously received SG in the parent study (IMMU-132-05) will continue to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until PD, toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
  Interventions: Drug: Sacituzumab Govitecan-hiy
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15) (Experimental): All participants who previously received SG in the parent study (IMMU-132-15) will continue to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until PD, toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
  Interventions: Drug: Sacituzumab Govitecan-hiy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hiy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132

SUMMARY:
The goal of this clinical study is to learn more about the study drug, sacituzumab govitecan-hziy (SG), and how safe it is in participants with metastatic cancer (cancer that has spread).

DETAILED DESCRIPTION:
This is a rollover study. Only participants who continue to receive clinical benefit from continuation of SG therapy and are tolerating therapy at the time of enrollment are eligible for this study. Participants enrolled may continue to receive SG at the dose that they were receiving in the Gilead parent study at the time of consenting to participate in this rollover study.

ELIGIBILITY:
Key Inclusion Criteria:

* Receiving ongoing treatment with sacituzumab govitecan in a Gilead (previously Immunomedics)-sponsored parent study.
* Continuing to receive clinical benefit from sacituzumab govitecan-hziy therapy.

Key Exclusion Criteria:

* Females who are pregnant or lactating.
* Initiated therapy with another cancer therapeutic agent since receiving last dose of study drug on the parent study in which they participated.
* Experienced a toxicity from sacituzumab govitecan-hziy that resulted in permanent discontinuation of therapy.
* Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (16):
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Christiana Care Health Services, Christiana Hospital, Newark, Delaware
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Baptist Health - Miami Cancer Institute, Miami, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - University of MD Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - New York Cancer & Blood Specialists - Setauket Medical Oncology, Port Jefferson, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Next Oncology, Austin, Texas
  - Oncology Consultants,P.A., Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - CHU UCL NAMUR - Sainte Elisabeth, Namur
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=IMMU-132-14

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Belgium and France.
Pre-assignment Details: 27 participants were screened. Participants must have been enrolled in other Gilead (previously Immunomedics)-sponsored studies of SG to be eligible to receive continued access to SG in this study.
Groups:
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01): All participants who previously received SG in the parent study (IMMU-132-01) continued to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until progressive disease (PD), toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05): All participants who previously received SG in the parent study (IMMU-132-05) continued to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until PD, toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
- Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15): All participants who previously received SG in the parent study (IMMU-132-15) continued to receive the same dose of SG up to a maximum of 10 mg/kg, on Days 1 and 8 of 21-day cycle until PD, toxicity, withdrawal of consent, lost to follow-up or loss of clinical benefit, or sponsor termination of the study was documented and were followed for long-term safety up to maximum 3.9 years.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15)
Started | 3 | 10 | 12
Completed | 0 | 0 | 0
Not Completed | 3 | 10 | 12
Not completed — Adverse Events Resolution or Stabilization | 3 | 4 | 0
Not completed — Death | 0 | 3 | 3
Not completed — Reason Not Specified | 0 | 2 | 4
Not completed — Withdrawal of Consent | 0 | 0 | 5
Not completed — Site Terminated by Sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Participants Analysis Set included all participants who received ≥ 1 dose of study drug following enrollment into this rollover IMMU-132-14 study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15) | Total
Number analyzed (Participants) | 3 | 10 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 8 | 10 | 18
  >=65 years | 3 | 2 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5.7) | 61 (10.4) | 49 (15.5) | 56 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 8 | 21
  Male | 0 | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 3 | 10 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 3 | 7 | 9 | 19
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 2 | 0 | 2
  United States | 3 | 7 | 12 | 22
  France | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a participant administered a medicinal product that does not necessarily have a causal relationship with this treatment.
Time Frame: First dose date up to 30 days post last dose (Up to 3.9 years)
Population: Participants from All Treated Participants Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15)
Number analyzed (Participants) | 3 | 10 | 12
percentage of participants | 66.7 | 100.0 | 91.7

2. Primary Outcome: Percentage of Participants Experiencing Any Serious Adverse Events
Description: A serious adverse event (SAE) was any untoward medical occurrence that, at any dose, was fatal (resulting in death), was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: First dose date up to 30 days post last dose (Up to 3.9 years)
Population: Participants from All Treated Participants Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15)
Number analyzed (Participants) | 3 | 10 | 12
percentage of participants | 0 | 40.0 | 8.3

3. Primary Outcome: Percentage of Participants Experiencing Any Grade and Grade 3 or 4 Laboratory Abnormalities
Description: The percentage of participants experiencing any clinically significant laboratory abnormality was summarized.
Time Frame: First dose date up to 30 days post last dose (Up to 3.9 years)
Population: Participants from All Treated Participants Analysis Set with at least 1 grade change postbaseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15)
Number analyzed (Participants) | 3 | 9 | 11
percentage of participants
  Any Grade 1 or Higher Laboratory Abnormalities | 100.0 | 88.9 | 81.8
  Grade 3 or 4 Laboratory Abnormalities | 33.3 | 44.4 | 72.7

ADVERSE EVENTS:
Time Frame: Up to 3.9 years
Description: All-Cause Mortality included all deaths occurred during study due to any cause among participants from All Treated Participants Analysis Set.
  Adverse Events included any serious or other (not including serious) AEs among All Treated Participants Analysis Set defined as all participants who received ≥ 1 dose of study drug following enrollment into this rollover IMMU-132-14 study.
Arm/Group | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15)
All-Cause Mortality (participants affected / at risk) | 0/3 | 3/10 | 3/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/10 | 1/12
Other Adverse Events (participants affected / at risk) | 2/3 | 10/10 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) (N=3) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) (N=10) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15) (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-01) (N=3) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-05) (N=10) | Sacituzumab Govitecan-hziy (Parent Study: IMMU-132-15) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 4
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 4 | 2
Gait disturbance (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Vaccination site pain (General disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 3 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Brain fog (Nervous system disorders) | 0 | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Paralysis (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Visuospatial deficit (Nervous system disorders) | 0 | 1 | 0
Device deposit issue (Product Issues) | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Iliac artery disease (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04319198/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04319198/SAP_001.pdf